CLINICAL TRIAL: NCT05770375
Title: Tolerability of MDMA in Schizophrenia
Acronym: TMS
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Anya Bershad, MD, PhD (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor-Investigator, Anya Bershad, MD, PhD, Principal Investigator, University of California, Los Angeles
Organization: University of California, Los Angeles (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB#22-001600; 1DP5OD036172-01 (NIH)
Record Dates: First submitted 2023-02-21; First posted 2023-03-15 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — N-Methyl-3,4-methylenedioxyamphetamine

STUDY DESIGN:
Intervention Model Description: Ascending-dose tolerability study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- MDMA (Experimental): Each subject will receive 3 doses of MDMA in ascending order: 40mg, 80mg, 120mg.
  Interventions: Drug: MDMA 40mg; Drug: MDMA 80mg; Drug: MDMA 120mg

INTERVENTIONS:
Drug: MDMA 40mg — MDMA 40mg
Drug: MDMA 80mg — MDMA 80mg
Drug: MDMA 120mg — MDMA 120mg

SUMMARY:
Impaired social motivation, or "asociality," is a negative symptom of schizophrenia (SCZ) and a cause of significant functional impairment in the illness. Whereas many symptoms of schizophrenia can be treated with antipsychotic medications, deficits in social motivation persist, leading to significant social disability in patients. There is currently no effective treatment for this symptom of the illness. One promising and unexplored avenue to enhance social motivation in schizophrenia is ± 3,4-methylenedioxymethamphetamine (MDMA). MDMA is a psychostimulant that shares some pharmacological properties with amphetamines, but in addition, has pronounced pro-social effects, increasing the motivation to engage socially. In healthy volunteers, it produces feelings of empathy and closeness with others and increases attention to positive social cues, perhaps partly through its effects on the social bonding hormone, oxytocin. MDMA has shown promise in other psychiatric conditions such as PTSD. Thus, MDMA could offer a unique therapeutic benefit in patients with SCZ who suffer from impaired social motivation. The investigators plan to take the first step in testing MDMA as a treatment for these social deficits by testing the tolerability of the drug in patients with SCZ. This will be an open-label, ascending-dose, within-subject trial in which participants will receive 40mg, 80mg, or 120mg of MDMA. The doses will be administered in ascending order, but doses will be stopped if subjects experience moderate or greater psychotic symptoms at 24 hours. This trial will assess the tolerability of the drug in this population and guide in the selection of a maximum well-tolerated dose for future studies. The primary tolerability measure will be clinician-rated psychotic symptoms (disorganized speech, delusions, hallucinations) collected at 24 hours after MDMA administration. The results of this project will lay the foundation for further investigations of MDMA and other psychoactive compounds as a treatment for debilitating and difficult-to-treat social deficits in schizophrenia. Future studies will examine interactions between the effects of psychoactive compounds and nonpharmacologic psychosocial interventions targeting social symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-60
* able to understand spoken English sufficiently to comprehend testing procedures
* DSM-5 diagnosis of schizophrenia, based on clinical interview
* clinical stability (i.e., no inpatient hospitalizations for six months prior to enrollment, no changes in medication in for 6 months prior to enrollment)

Exclusion Criteria:

* no history of aggressive or suicidal behavior while psychotic
* no history of IQ less than 70 or developmental disability, based on medical history
* no clinically significant neurological disease (e.g., epilepsy), or cardiovascular condition (e.g. cardiac arrhythmia) based on medical history
* no history of serious head injury (i.e., loss of consciousness longer than 1 hour, neuropsychological sequelae, cognitive rehabilitation treatment after head injury) based on medical history
* no substance or alcohol use disorder in the past six months
* no sedatives or benzodiazepines within 24 hours of testing
* no positive urine toxicology screen or visible intoxication on the day of assessment
* no women who are pregnant or think that they might be pregnant, based on self-report and urine test
* not currently taking SSRIs or SNRIs
* no history of NMS or serotonin syndrome
* No prolongation of the QTc interval on EKG

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Positive and Negative Syndrome Scale for Schizophrenia (PANSS): Disorganized speech. | 24 hours after each drug session
  The PANSS is a validated 30-item clinician-administered scale assessing symptom severity in SCZ. It is widely used to assess the efficacy of antipsychotic medications. Symptoms are rated from 1 (not present) to 7 (extremely severe). The PANSS will be administered at the first session, before drug administration at each drug session, and 24 hours after each drug session. Our primary tolerability outcome measure will be clinician-rated psychotic symptoms on the three core DSM-V symptoms of psychosis (disorganized speech, delusions, hallucinations) on the PANSS 24 hours after each drug session. This is the item assessing disorganized speech.
Positive and Negative Syndrome Scale for Schizophrenia (PANSS): Delusions | 24 hours after each drug session
  The PANSS is a validated 30-item clinician-administered scale assessing symptom severity in SCZ. It is widely used to assess the efficacy of antipsychotic medications. Symptoms are rated from 1 (not present) to 7 (extremely severe). The PANSS will be administered at the first session, before drug administration at each drug session, and 24 hours after each drug session. Our primary tolerability outcome measure will be clinician-rated psychotic symptoms on the three core DSM-V symptoms of psychosis (disorganized speech, delusions, hallucinations) on the PANSS 24 hours after each drug session. This is the item assessing delusions.
Positive and Negative Syndrome Scale for Schizophrenia (PANSS): Hallucinations | 24 hours after each drug session
  The PANSS is a validated 30-item clinician-administered scale assessing symptom severity in SCZ. It is widely used to assess the efficacy of antipsychotic medications. Symptoms are rated from 1 (not present) to 7 (extremely severe). The PANSS will be administered at the first session, before drug administration at each drug session, and 24 hours after each drug session. Our primary tolerability outcome measure will be clinician-rated psychotic symptoms on the three core DSM-V symptoms of psychosis (disorganized speech, delusions, hallucinations) on the PANSS 24 hours after each drug session. This is the item assessing hallucinations.

CONTACTS AND LOCATIONS:
Locations (1):
- UCLA, Los Angeles, California, United States